CLINICAL TRIAL: NCT02953860
Title: Phase II Trial of Fulvestrant Plus Enzalutamide in ER+/Her2- Advanced Breast Cancer
Brief Title: Fulvestrant Plus Enzalutamide in ER+/Her2- Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1001.cc
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: Advanced Breast Cancer; ER+/Her2 Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fulvestrant with Enzalutamide (Experimental): 500mg of Fulvestrant will be given IM on days 1, 15, 28, then every 4 weeks as per standard of care (SOC) and 160mg of Enzalutamide will be given, in conjunction with Fulvestrant, PO daily.
  Interventions: Drug: Fulvestrant with Enzalutamide

INTERVENTIONS:
Drug: Fulvestrant with Enzalutamide — 500mg of Fulvestrant will be given IM on days 1, 15, 28, then every 4 weeks as per standard of care (SOC) and 160mg of Enzalutamide will be given PO daily. Patients will receive a tumor biopsy at the start of treatment and 4 weeks after the start of treatment, with an optional 3rd biopsy at the end treatment.
  Other Names: FASLODEX; MDV3100

SUMMARY:
A phase 2 study to evaluate the tolerability and clinical activity of adding enzalutamide to fulvestrant treatment in women with advanced breast cancer that are ER and/or PR positive and Her2 normal.

DETAILED DESCRIPTION:
This is a single arm, non-randomized, open-label phase 2 study designed to evaluate the tolerability and clinical activity of adding enzalutamide to fulvestrant treatment in women with advanced breast cancer that are ER and/or PR-positive and Her2 normal. In this study 500 mg of Fulvestrant will be given IM on days 1, 15, 28, then every 4 weeks as per standard of care (SOC) and 160mg of Enzalutamide will be, in conjunction with Fulvestrant, PO daily.

ELIGIBILITY:
Inclusion Criteria:

1. ER+ Her2- breast cancer
2. Metastatic
3. Female, at least 18 years of age
4. Candidate for fulvestrant therapy - patients who have started fulvestrant may enter this trial if within 3 months of starting fulvestrant
5. Measurable or evaluable by RECIST 1.1
6. ECOG PS 0-2
7. Able to swallow study drug and comply with study requirements
8. Tumor available for fresh biopsy (two biopsies - pretreatment as regards enzalutamide, and during treatment at 4 weeks). The patient will be also be asked if they would be willing to provide a third biopsy at time of progression.
9. If patient is pre- or peri- menopausal, then will need to have concurrent ovarian suppression. Patients may have already gotten the loading dose of ovarian suppression. Pre- or peri- menopausal subjects must have a negative urine pregnancy test confirmed at screening.
10. ANC >1000/uL and platelets >75,000/uL at screening visit
11. Total bilirubin < 1.5 times upper limit of normal (ULN) at the screening visit unless an alternate nonmalignant etiology exists (eg, Gilbert's disease)
12. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 times ULN or < 5 times ULN if patient has documented liver metastases
13. Creatinine < 1.5 times ULN
14. INR < 1.5 times ULN, or if on warfarin, can safely transition off for biopsy
15. Willing to donate blood for research at 4 time points
16. Written informed consent obtained prior to biopsies and blood samples
17. Agreement to exercise appropriate use of contraception. Subjects should use 2 acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at the time of screening for an enzalutamide study and continuing throughout the course of treatment and for at least three months after enzalutamide is discontinued.

Exclusion Criteria:

1. Current or previously treated brain or leptomeningeal metastases
2. History of seizures
3. Prior treatment with an anti-androgen (abiraterone, ARN-509, bicalutamide, enzalutamide, ODM-201, TAK-448, TAK-683, TAK-700, VT-464)
4. Systemic estrogens or androgens within 14 days before initiating therapy. Vaginal estrogens are allowed if necessary for patient comfort.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2020-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D Elias, MD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado, Aurora, Colorado
  - Lone Tree Medical Center, Lone Tree, Colorado
  - West Cancer Center, Germantown, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fulvestrant With Enzalutamide
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: age 18 and up
Arm/Group | Fulvestrant With Enzalutamide
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 61 [46 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 27
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate of the Combination of Enzalutamide/ Fulvestrant
Description: To determine the clinical benefit rate at 24 weeks of the combination of enzalutamide/fulvestrant. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT scan or by caliper. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR; clinical benefit rate (CBR) at 24 weeks (CR + PR + stable disease lasting at least 24 weeks.
Time Frame: 24 Weeks
Population: All eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant With Enzalutamide
Number analyzed (Participants) | 32
Participants | 7

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Safety Profile)
Description: The safety of the combination of enzalutamide with fulvestrant will be assessed according to CTCAE 4.03.
Time Frame: 24 Weeks
Population: all eligible patients
Measure: Number; unit: participants
Arm/Group | Fulvestrant With Enzalutamide
Number analyzed (Participants) | 32
participants
  fatigue | 17
  nausea | 16
  vomiting | 9
  constipation | 10
  headache | 11
  diarrhea | 7
  cognitive dysfunction | 5

3. Secondary Outcome: Percent Progression Free at 24 Weeks
Description: PFS is defined as the time from the first day of enzalutamide treatment (Study Day 1) until documented disease progression or death on study, whichever occurs first. Percent (%) progression free at 24 weeks is the number of patients without disease progression after 24 weeks follow-up.
Time Frame: Up to 24 Weeks
Population: all eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant With Enzalutamide
Number analyzed (Participants) | 32
Participants | 7

ADVERSE EVENTS:
Time Frame: AEs collected during treatment (which lasted up to a year)
Description: CTCAE 4.0 Collected with each monthly visit, patients kept diary.
Arm/Group | Fulvestrant With Enzalutamide
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 2/32
Other Adverse Events (participants affected / at risk) | 17/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant With Enzalutamide (N=32)
myocardial infarction (Cardiac disorders) | 1 (1) — Felt not to be related to treatment. Unrelated to fulvestrant unlikely related to enzalutamide
cholecystitis (Hepatobiliary disorders) | 1 (1) — unrelated to fulvestrant and enzalutamide
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant With Enzalutamide (N=32)
Fatigue (General disorders) | 17 (17)
Hot Flashes (Endocrine disorders) | 6 (6)
insomnia (Nervous system disorders) | 6 (6)
nausea (Gastrointestinal disorders) | 16 (16)
vomiting (Gastrointestinal disorders) | 9 (9)
constipation (Gastrointestinal disorders) | 10 (10)
anorexia (Gastrointestinal disorders) | 9 (9)
headache (Nervous system disorders) | 11 (11)
achiness (Musculoskeletal and connective tissue disorders) | 14 (14)
cognitive dysfunction (Nervous system disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
limited size of trial not randomized heavily pretreated somewhat heterogeneous population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT02953860/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT02953860/ICF_001.pdf